CLINICAL TRIAL: NCT03053804
Title: Clinical Application of MR-PET in Non-small Cell Lung Cancer: Diagnosis, Treatment, Outcome, and Prognosis Prediction
Brief Title: Clinical Application of MR-PET in Non-small Cell Lung Cancer: Diagnosis, Treatment Outcome, and Prognosis Prediction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201501073RINA
Record Dates: First submitted 2016-10-30; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2016-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: MR/PET; Non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MR/PET (Experimental): hypothesize that MR/PET can have better information than current CT image study
  Interventions: Radiation: MR/PET

INTERVENTIONS:
Radiation: MR/PET — MR/PET with contrast media and FDG-18

SUMMARY:
It is a study that hypothesize that MR/PET can have better information than current CT image study, about the medical or surgical treatment outcome of lung cancer

DETAILED DESCRIPTION:
The investigators analyze tumor size、ADCmean、ADCmin、DCE、SUVmax、SUVmin、etc in MR/PET study，to compare its efficacy with other image studies in tumor malignancy grade, systemic involvement detection, treatment outcome after medical target therapy and treatment outcome after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 20 years old.
2. Patients have confirmed lung cancer by histopathological methods (fiber, bronchoscopy, lung biopsy, open chest biopsy, pleural effusion exfoliated cells, sputum exfoliated cells)
3. Patients voluntarily to join this study and signed informed consents.

Exclusion Criteria:

1. Any body metal implants (pacemaker implantation, nerve stimulator, vascular stent, aneurysm clip, eye foreign body, the inner metal prosthesis) or artificial heart valves
2. Patients with claustrophobia to MRI examination
3. Patients who are reluctant to comply with follow-up and subsequent examination
4. The other condition that do not meet the inclusion criteria.
5. Pregnancy.
6. Age < 20 years old.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline PET/MR parameters at 2 months after treatment | 2 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yeun-Chung Chang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No